CLINICAL TRIAL: NCT06780566
Title: Routine Application of Point-of-care PCR Test to Identify and Direct Therapy for Acute Respiratory Infection in the Emergency Department (RAPID-ARIED) Trial
Brief Title: Routine Application of Point-of-care PCR Test to Identify and Direct Therapy for Acute Respiratory Infection in the Emergency Department Trial
Acronym: RAPID-ARIED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lam Pui Kin, Clinical Associate Professor of Practice, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RAPID-ARIED1
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Influenza; COVID-19; Acute Respiratory Infections (ARIs)
Keywords: COVID-19; Acute respiratory infections; Point-of-care testing; Polymerase Chain Reaction; Randomized controlled trial; emergency department; Influenza
MeSH Terms: conditions — Influenza, Human; COVID-19; Emergencies

STUDY DESIGN:
Intervention Model Description: After obtaining informed consent, each recruited participant will be given a unique participant identification number. Research team members will then use this identification number to randomise participants in a 1:1 ratio to either the intervention group or the control group. Permuted blocks of varying size (4, 6, and 8) will be generated using internet-based randomisation software
Masking Description: Not applicable because this is an open-label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Point-of-care PCR testing for respiratory viruses in the ED
  Interventions: Diagnostic Test: Point-of-care PCR testing for respiratory viruses
- Control Group (Other): Laboratory PCR testing for respiratory viruses after admission to the hospital floor
  Interventions: Diagnostic Test: Laboratory PCR testing for respiratory viruses

INTERVENTIONS:
Diagnostic Test: Point-of-care PCR testing for respiratory viruses — A nasal swab will be collected by trained research staff in full personal protective equipment (PPE) and placed into 3 mL of viral transport medium. The sample will be immediately processed and analysed in the ED using the Xpert® Xpress SARS-CoV-2/Flu/RSV test according to the manufacturer's instructions. The results of the test will be documented in the patient's paper or electronic case notes, and the clinical team will be directly informed of all results. The participant or legal guardian who signs the consent form will also be informed of the results when appropriate.
  Arms: Intervention Group
Diagnostic Test: Laboratory PCR testing for respiratory viruses — The ordering of test for respiratory pathogens will be decided by the treating clinical team. All tests will be performed using the standard methods of the hospital laboratory.
  Arms: Control Group

SUMMARY:
The RAPID-ARIED Trial is a pragmatic, single-centre, parallel group, open-label, randomised controlled trial to be conducted in the Accident and Emergency Department of Queen Mary Hospital in Hong Kong. The investigators aim to 1) to evaluate the clinical impact of the routine application of point-of-care polymerase chain reaction (PCR) testing for targeted respiratory pathogens in the emergency department (ED) for adult patients with acute respiratory infections (ARIs) on the hospital length of stay (LOS), antiviral and antibiotic use during influenza seasons or future waves of COVID-19; and 2) to conduct a health economic analysis of such a strategy.

The investigators hypothesise that in adult patients hospitalised from the ED for ARIs during influenza seasons or COVID-19 waves, routine point-of-care PCR test for influenza A&B, SARS-CoV-2 and respiratory syncytial virus in the ED reduces the hospital LOS significantly and cost effectively compared to usual care.

In total, 1,050 adult patients who are intended to be admitted to hospital with ARIs in the ED will be recruited during influenza seasons or future waves of COVID-19 over 36 months from 2025 to 2027.

Participants will be randomised (1:1 ratio) into the interventional group and control group. A nasal swab will be collected. In the intervention group, research staff will perform PCR test using the GeneXpert® Xpress PCR kit in the ED and communicate the test results to the patient and the clinical team. In the control group, all microbiology tests will be determined by the clinical team, with retrospective PCR testing of the nasal swab sample after 28 days.

The primary outcome is the median hospital LOS. Secondary outcomes include antivirals and antibiotics use and administration time, mortality, and quality-adjusted life year, assessed using the EQ-5D-5L questionnaire.

Intention-to-treat analysis (superiority framework) and cost-effectiveness analysis (from healthcare provider perspective) will be conducted.

Study results will provide evidence regarding the optimal PCR testing strategy in the future influenza seasons and COVID-19 waves.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or above
* Intended for admission to hospital with acute respiratory illness (defined as a provisional diagnosis of pneumonia, bronchitis, influenza-like illness, acute exacerbation of chronic obstructive pulmonary disease, asthma or bronchiectasis.)
* Respiratory symptoms present ≤10 days before admission to hospital
* No prior treatment with antibiotics or antivirals in the previous 14 days

Exclusion Criteria:

* Refusal of nasal or pharyngeal swabbing
* Refusal of informed consent
* Previously included in the study and re-presentation within 28 days of hospital discharge
* A prior positive test by antigen test or other PCR test for COVID-19 or influenza before ED presentation
* Exposure to FluMist® or other similar live attenuated influenza vaccines within 1 month (because such exposures may lead to a false positive PCR test result with the nasal swab sample).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | From enrollment to day 28
  Hospital length of stay in days

SECONDARY OUTCOMES:
Neuraminidase inhibitors use | From enrollment to day 28
  Proportion of neuraminidase inhibitor use in patients with and without influenza
Nirmatrelvir-ritonavir or molnupiravir use | From enrollment to day 28
  Proportion of nirmatrelvir-ritonavir or molnupiravir use in patients with and without COVID-19
Median time to antiviral commencement from ED registration | From enrollment to day 28
  Median time to antiviral commencement from ED registration in hours
Antibiotic use | From enrollment to day 28
  Proportion of antibiotic use in patients
Median time to antibiotic commencement from ED registration | From enrollment to day 28
  Median time to antibiotic commencement from ED registration in hours
ICU admission | From enrollment to day 28
  Proportion of patients requiring admission to an intensive care unit (ICU) or a high dependency unit (HDU), censored at 28 days post-enrolment
ICU length of stay | From enrollment to day 28
  Median duration of stay in ICU and/or HDU in days
Proportion of patients requiring non-invasive ventilation during their hospital stay | From enrollment to day 28
  Proportion of patients requiring non-invasive ventilation during their hospital stay
Proportion of patients requiring mechanical ventilation during their hospital stay | From enrollment to day 28
  Proportion of patients requiring mechanical ventilation during their hospital stay
Ventilator-free days | From enrollment to day 28
  Ventilator-free days
28-day All-cause mortality | From enrollment to day 28
  All-cause mortality
In-hospital mortality | From enrollment to day 28
  In-hospital mortality
Proportion of patients readmitted to hospital within 28 days of hospital discharge | From hospital discharge to day 28 after hospital discharge
  Proportion of patients readmitted to hospital within 28 days of hospital discharge
Health-related quality of life | Day 1 ,7, 14, 28
  Health-related quality of life measured with five-level EuroQol five-dimensional questionnaire (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Pui Kin Rex Lam, MBBS, MPH, FHKCEM, Principal Investigator — The University of Hong Kong
Locations (1):
- Accident and Emergency Department, Queen Mary Hospital, Hong Kong, None Selected, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
IPD requires additional IRB approval because of local patient privacy ordinance.